CLINICAL TRIAL: NCT07250347
Title: Langue and Imaging-integrated Foundation Model for Gastric Cancer Detection and Staging Via Contrast-Enhanced CT: a Multicenter Study
Brief Title: AI-Assisted Detection and Staging of Gastric Cancer Using Contrast-Enhanced CT
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Jiangsu Cancer Institute & Hospital (Other); The Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital (Unknown); Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-SR-842
Record Dates: First submitted 2025-09-29; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Gastric Cancer Stage; Gastric Cancer Patients Undergoing Gastrectomy
Keywords: Gastric cancer; stage; artificial-intelligence; detection; contrast-enhanced CT
MeSH Terms: conditions — Stomach Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1 (Internal Derivation Cohort): Retrospective case-only cohort of adults with pathologically confirmed gastric cancer who underwent preoperative contrast-enhanced CT at the sponsoring institution. Existing CT images and clinical/pathology records will be used to train and test the AI model and to estimate diagnostic performance for T and N staging.
  Interventions: Diagnostic Test: CT scan
- Cohort 2 (External Validation Cohort A): Independent retrospective case-only cohort from an external hospital with the same inclusion/exclusion criteria. Used solely for external validation to assess reproducibility across sites and scanners.
  Interventions: Diagnostic Test: CT scan
- Cohort 3 (External Validation Cohort B): A second independent retrospective validation cohort from another institution to further test generalizability.
  Interventions: Diagnostic Test: CT scan

INTERVENTIONS:
Diagnostic Test: CT scan — preoperative contrast-enhanced CT

SUMMARY:
Accurate preoperative assessment of gastric cancer stage guides eligibility for endoscopic resection, extent of gastrectomy and lymphadenectomy, selection for neoadjuvant therapy, and use of staging laparoscopy. Contrast-enhanced CT (CECT) is guideline-endorsed for initial staging, yet performance varies across institutions and readers. This study will evaluate an artificial-intelligence (AI) system that analyzes routine CECT to detect gastric cancer and assign four-class T stage (T1-T4) and N stage (N0-N3) .

DETAILED DESCRIPTION:
Adults with confirmed gastric cancer undergoing pre-treatment CECT will be enrolled. The AI analysis will be applied to clinically acquired images. Radiologist interpretations with and without AI support will be collected in a prespecified reader study. The reference standard will include surgical pathology, supplemented by clinical follow-up when applicable. The primary outcome is detection performance, diagnostic performance of the AI for four-class staging (e.g., accuracy and area under the receiver operating characteristic curve). Secondary outcomes include the effect of AI assistance on reader accuracy and interpretation time, inter-reader agreement, and cross-site reproducibility.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically confirmed gastric cancer;
2. preoperative contrast-enhanced CT performed;
3. no evidence of distant metastasis on baseline staging;
4. curative-intent management with complete postoperative histopathology.

Exclusion Criteria:

1. prior treatment before surgery;
2. non-diagnostic or poor-quality CT precluding evaluation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll adult patients (≥18 years old) with a confirmed diagnosis of gastric cancer (adenocarcinoma) who have undergone contrast-enhanced CT (CECT) as part of their standard preoperative evaluation. Participants will be selected from both internal and external cohorts, with inclusion from multiple centers to assess cross-site reproducibility and generalizability of the AI model.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of the AI model for staging | 3 years
  The primary outcome is the diagnostic accuracy of the AI system for four-class T staging (T1-T4) and N staging (N0-3) based on contrast-enhanced CT. The AI performance will be assessed using accuracy, area under the receiver operating characteristic curve (AUC), and micro-AUC for internal and external cohorts.

SECONDARY OUTCOMES:
Reader Accuracy with AI Support | 3 years
  This outcome measures the accuracy of radiologists in classifying gastric cancer stagewhen aided by the AI system compared to manual classification without AI assistance. Accuracy will be compared between different radiologist experience levels.
Survival time | 3 years
  Calculate the survival time of gastric cancer patients from the point of diagnosis and treatment initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Yudong, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No